CLINICAL TRIAL: NCT05154656
Title: Fast Three-Dimensional Black Blood Magnetization Prepared Spiral Fast Spin Echo T1rho Relaxometry for Early Diagnosis of Liver Fibrosis
Brief Title: Three-Dimensional T1rho Using Spiral Fast Spin Echo
Status: Withdrawn | Type: Observational
Why Stopped: We did not get the grant support.
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chen Weitian, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2018.611
Record Dates: First submitted 2021-12-09; First posted 2021-12-13 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Liver Fibrosis
Keywords: 3D, T1rho, Fast spin echo
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with early stage of liver fibrosis
- subjects with no liver fibrosis

SUMMARY:
Liver fibrosis is the main feature in early chronic liver diseases. If identified early, liver fibrosis is reversible. The current gold standard for diagnosing liver fibrosis is invasive liver biopsy. Existing non-invasive methods still have significant limitations.

T1rho imaging is a promising non-invasive technology evaluating liver fibrosis. It does not require exogenous contrast agent or extra hardware. However, it remains challenging to perform T1rho measurements of the liver. The rich blood signal in the liver introduces quantification errors of liver parenchyma. The existing black blood MRI technologies are based on Cartesian FSE acquisitions, which are not optimal for liver imaging. The residual blood signal is often observed which confounds the measurement. Current T1rho measurement of the liver is mostly performed in two-dimension. 3D coverage of liver is desirable. However, 3D T1rho imaging of liver suffers from long scan time due to increased spatial coverage, reduced scan time efficiency from motion compensation, and high specific absorption rate (SAR).

The investigators aim to overcome these challenges by developing 3D T1rho imaging technologies based on magnetization prepared spiral FSE acquisition. Compared to Cartesian FSE, Spiral FSE traverses k-space more efficiently per unit of time, and has reduced SAR due to significantly decreased number of radiofrequency pulses in the echo trains. Spiral acquisition has zero gradient moment at the kspace center, which substantially reduces its sensitivity to respiratory motion. The residual motion manifests as benign incoherent artifacts in the image domain rather than detrimental structured artifacts. Differently to Cartesian FSE, Spiral FSE provides flexibility to design and optimize flow-sensitizing gradients throughout the echo trains to achieve superior suppression of blood signal. The investigators will evaluate the proposed pulse sequences in both healthy controls and patients with liver fibrosis.

This project will provide new black blood imaging technologies and a 3D diagnostic tool for early detection of liver fibrosis. This will improve clinical outcomes for patients with chronic liver disease, and provide a springboard for further development of MRI technology for other purposes.

ELIGIBILITY:
Inclusion Criteria:

* Between age 18 and age 55
* patients with early liver fibrosis
* Informed written consent obtained

Exclusion Criteria:

* Contraindications to MRI such as the presence of metallic implants, claustrophobia and pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 60 patients with early stage of liver fibrosis and 60 subjects with no liver fibrosis
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Analysis of variance (ANOVA) will be performed to compare the measurement between subjects with no fibrosis and subjects with early stage fibrosis | one year
  Correlations will be calculated to assess the correlation between the disease state determined by histology and the imaging measurements

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Prince of Wale Hospital, Hong Kong, Shatin, Hong Kong